CLINICAL TRIAL: NCT03660436
Title: An Open-label, Single-sequence Study to Investigate the Effects of BMS-986165 at Steady State on the Single Dose Pharmacokinetics of Mycophenolate Mofetil (MMF) in Healthy Male Subjects
Brief Title: An Investigational Study of Experimental Medication BMS-986165 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-071
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986165 + MMF (Experimental): Oral administration
  Interventions: Drug: BMS-986165; Drug: MMF

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
Drug: MMF — Specified dose on specified days
  Other Names: Mycophenolate Mofetil

SUMMARY:
The purpose of this study is to investigate the effects of experimental medication BMS-986165 in healthy male participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participant, as determined by no clinically significant deviation from normal in physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body mass index of 18.0 to 32.0 kg/m2, inclusive, and weight ≥ 50 kg, at screening
* Normal renal function at screening as evidenced by an estimated GFR (glomerular filtration rate) > 80 mL/min/1.732 m2

Exclusion Criteria:

* Any medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease
* Positive anti- John Cunningham virus (JCV) antibody test at Screening
* History of allergy to MMF, BMS-986165, related compounds or any significant drug allergy

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of mycophenolic acid (MPA) | 18 days
Area under the concentration vs time curve from time zero to the last quantifiable plasma concentration (AUC[0-T]) of MPA | 18 days
AUC extrapolated to infinity (AUC[INF]) of MPA | 18 days

SECONDARY OUTCOMES:
Number of adverse events (AE) | Up to 48 days
Number of serious adverse events (SAE) | Up to 48 days
Number of AEs leading to discontinuation | Up to 48 days
Incidence of clinically significant changes in laboratory test results, vital sign measurements, electrocardiograms (ECGs) and physical examination results | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm